CLINICAL TRIAL: NCT03439020
Title: The Efficacy of a Fully Covered Self-expandable Metal Stent Anchored by a Plastic Stent for Anti-migration in the Management of Malignant Biliary Strictures: a Prospective Randomized Controlled Study
Brief Title: The Efficacy of Plastic Stent Anchoring to Reduce Migration of Metal Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1709-081-886
Record Dates: First submitted 2018-02-01; First posted 2018-02-20 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Malignant Biliary Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCSEMS + Plastic (Experimental): Insert a fully covered self expandable metal stent (FCSEMS) for malignant biliary stricture and insert an additional plastic stent to anchor the metal stent.
  (Plastic stent anchoring)
  Interventions: Procedure: Plastic stent anchoring; Procedure: FCSEMS
- FCSEMS (Active Comparator): Insert only a fully covered self expandable metal stent (FCSEMS) without a plastic stent for malignant biliary stricture.
  Interventions: Procedure: FCSEMS

INTERVENTIONS:
Procedure: Plastic stent anchoring — Insert an additional plastic stent to anchor the fully covered self expandable metal stent.
  Arms: FCSEMS + Plastic
Procedure: FCSEMS — Insert a fully covered self expandable metal stent (FCSEMS) for malignant biliary stricture

SUMMARY:
The aim of this study is to demonstrate that the group with an additional plastic stent to anchor the fully covered self expandable metal stent (FCSEMS) in patients with malignant biliary stricture has less stent migration than the group with FCSEMS only. The primary outcome is stent migration for 6 months. The secondary outcomes are stent related adverse events, stent patency, and overall survival.

DETAILED DESCRIPTION:
Endoscopic retrograde biliary drainage using a plastic stent for the treatment of malignant biliary stricture has advantages in that it is easy to perform and low cost, but it has a short period of patency. To overcome this drawback, self-expandable metal stents (SEMS) have been developed and are now widely used. But, over time, the SEMS also develop restenosis, due to tumor ingrowth and the tissue hyperplasia caused by the stimulation of the surrounding tissues by the metal thin wire. To overcome these disadvantages, a fully covered self-expandable metal stents (FCSEMS) covered with a polymer coating have been developed and used. However, the FCSEMS showed more stent migration than the uncovered SEMS, which was not superior to the uncovered SEMS in terms of loss of stent function. In order to overcome the limitations of the FCSEMS, small-scale studies have shown that stent migration can be reduced by anchoring the FCSEMS using a plastic stent. To date, there has been no randomized controlled study to determine whether the FCSEMS can be anchored with a plastic stent in patients with malignant biliary stricture to reduce the stent migration. Therefore, the purpose of this study is to evaluate the efficacy of plastic stent anchoring to reduce migration of FCSEMS.

ELIGIBILITY:
Inclusion Criteria:

* Malignant biliary stricture requiring biliary drainage through endoscopic procedure

Exclusion Criteria:

* Previous history of metal stent placement for malignant biliary stricture
* Hilar cholangiocarcinoma
* Malignant biliary stricture of intrahepatic duct
* A recurrence after surgery due to malignant biliary stricture
* Life expectancy less than 3 months
* Pregnancy
* If endoscopy is not possible based on the judgement of the researcher

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Stent migration rate | 6 months after randomization
  Stent migration is classified as proximal or distal migration. Proximal stent migration is defined as any migration of the FCSEMS(Fully covered self expandable metal stent) into the bile duct, preventing its easy removal.
  Distal stent migration is defined in three ways. The first is when the stent is completely distally migrated without being lodged into the duodenum.
  The second is when the stent is lodged in the distal bile duct below the stricture.
  The third case is when the stent is migrated to the distal portion of the stricture and is lodged in the duodenum opposite the papilla

SECONDARY OUTCOMES:
Stent-related adverse events | 6 months after randomization
  According to lexicon for endoscopic adverse events
Duration of stent patency | 6 months after randomization
  The period from the insertion of the stent to the point at which stent revision is required
Overall survival | 6 months after randomization
  Period from stenting to death

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Paik WH, Woo SM, Chun JW, Song BJ, Lee WJ, Ahn DW, Lee YS, Choi YH, Ryu JK, Kim YT, Lee SH. Efficacy of an internal anchoring plastic stent to prevent migration of a fully covered metal stent in malignant distal biliary strictures: a randomized controlled study. Endoscopy. 2021 Jun;53(6):578-585. doi: 10.1055/a-1256-0571. Epub 2020 Oct 8. PMID 32886935